CLINICAL TRIAL: NCT07267975
Title: Effectiveness of Intermittent Oral Iron Therapy vs Continuous Oral Iron Therapy in Treating Iron Deficiency Anemia Patients UpTo 5 Year of Age; a Randomized Control Trial
Brief Title: Effectiveness of Oral Iron Therapy in Iron Deficiency Anemia With Daily vs Alternate Day Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Marryam Kaleem, PGR, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No/1032/CH-UCHS
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-01

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency Anemia Treatment
Keywords: IDA, children, oral iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous oral iron therapy (Active Comparator): Oral iron daily dosing 6mg/kg/day
  Interventions: Drug: Ferrous sulphate
- Intermittent oral iron (Experimental): Oral iron therapy on alternate day with dose of 6mg /kg/day for 3 mons
  Interventions: Drug: Ferrous sulphate

INTERVENTIONS:
Drug: Ferrous sulphate — Continuous vs intermittent oral iron therapy to see the difference of Hemoglobin rose in both group
  Other Names: Daily dosing
  Arms: Continuous oral iron therapy
Drug: Ferrous sulphate — Pattern of Rise in hemoglobin in alternate day doaung
  Other Names: Intermittent, alternate day dosing
  Arms: Intermittent oral iron

SUMMARY:
Treating iron deficiency anemia in children with daily and alternate day oral iron therapy

DETAILED DESCRIPTION:
Comparison of effectiveness of oral iron in daily and alternate group in children

ELIGIBILITY:
Inclusion Criteria:

- Patients of both genders with ages in the range of 0 -60 months suffering from IDA as per operational definition.

Exclusion Criteria:

* Who have already taken treatment for IDA during last 2-months as per history/clinical record.

Who have undergone recent blood transfusion during last 12-weeks as per history/clinical record.

Children with chronic kidney disease, chronic liver disease, cardiac failure or concomitant malignancy

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Rise in hemoglobin level after oral iron | 3 months
  Hemoglobin level change in g/dl
Change in Hemoglobin level | 3month
  Hb rise in g/dl

SECONDARY OUTCOMES:
Rise in ferritin level | 3 month
  Ferritin level change in ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- University of child health science and the children hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Confidentiality